CLINICAL TRIAL: NCT06062446
Title: A Prospective, Single-Arm Study of a Modified Lumbar Puncture (LP) Procedure That Reduces Post-Lumbar Puncture Headaches (PLPH) in Adult Patients
Brief Title: A Prospective Study of a Modified Lumbar Puncture (LP) Procedure That Reduces Post-Lumbar Puncture Headaches (PLPH) in Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jay-Jiguang Zhu, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0732
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Post-Lumbar Puncture Headache
Keywords: lumbar puncture; headache
MeSH Terms: conditions — Post-Dural Puncture Headache; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Modified Lumbar Puncture (Experimental)
  Interventions: Procedure: Modified Lumbar Puncture

INTERVENTIONS:
Procedure: Modified Lumbar Puncture — The Investigator will perform the modified LP procedure using the 22 Gg needles Quincke spinal needle (namely, without reinsertion of stylet into the spinal needle after cerebrospinal fluid (CSF) collection before spinal needle removal).

SUMMARY:
The purpose of this study is to o determine whether the modified LP procedure reduces the incidence of PLPH to 5% or lower, to determine whether the modified LP procedure reduces the frequency of epidural blood patch (EBP) usage to 10% or lower of the PLPH population and to identify factors that may contribute to or reduce incidence of PLPH

ELIGIBILITY:
Inclusion Criteria:

* Participants who can sign informed consent
* Participants who have stated willingness to comply with all study procedures and availability for the duration of the study
* Participants receiving a LP per standard of care (SOC) need for diagnostic or therapeutic purposes only
* Participants with Karnofsky Performance Scale (KPS) ≥ 60

Exclusion Criteria:

* Participants with a past medical history of chronic headaches (≥15 days per month) or acute headaches
* Participants with recent neurosurgical device implants such as ventriculoperitoneal shunt
* Participants with more than one dural puncture during the same LP procedure
* Participants have chronic coagulopathy with elevated prothrombin time (PT), Partial thromboplastin time (PTT), and International Normalized ration (INR).
* Participants who are on active anticoagulant or antiplatelet therapy unless stopped such therapy prior to LP per SOC guidance.
* Participants with suspicions of raised intracranial pressure by either clinical assessment or imaging assessment or both
* Participants with severe spinal column deformities, such as scoliosis. Disc diseases are not exclusion criteria
* Participants with LP procedural complications that require a needle type or needle size change

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with headaches as assessed by a questionnaire | 30-60 minutes after LP
  Participants will answer "Yes" or "No" in response to 1-2 questions: 1) Do you have a headache? 2) If you answered "Yes" to the previous question, does the headache get better when you sit up?
Number of participants with headaches as assessed by a questionnaire | 1 day after LP
  Participants will answer "Yes" or "No" in response to 1-2 questions: 1) Do you have a headache? Or have you had a headache since the lumbar puncture? 2) If you answered "Yes" to the previous question, does the headache get better when you sit up?
Number of participants with headaches as assessed by a questionnaire | 3 days after LP
  Participants will answer "Yes" or "No" in response to 1-2 questions: 1) Do you have a headache? Or have you had a headache since the lumbar puncture? 2) If you answered "Yes" to the previous question, does the headache get better when you sit up?
Number of participants with headaches as assessed by a questionnaire | 5 days after LP
  Participants will answer "Yes" or "No" in response to 1-2 questions: 1) Do you have a headache? Or have you had a headache since the lumbar puncture? 2) If you answered "Yes" to the previous question, does the headache get better when you sit up?

SECONDARY OUTCOMES:
Number of participants that use the epidural blood patch | 1 day after the LP
Number of participants that use the epidural blood patch | 3 days after the LP
Number of participants that use the epidural blood patch | 5 days after the LP

CONTACTS AND LOCATIONS:
Overall Officials: Jay-Jiguang Zhu, MD,PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No